CLINICAL TRIAL: NCT05929092
Title: Total Body Irradiation/ Fludarabine/ Busulfan/ Cyclophosphamide (TFBC) Combined With Umbilical Cord Blood Transplantation (UCBT) in the Treatment of High-risk Malignant Hematological Diseases
Brief Title: TFBC Combined With UCBT in the Treatment of High-risk Malignant Hematological Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOOCHOW-WXJ-2023-132
Record Dates: First submitted 2023-06-24; First posted 2023-07-03 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Hematopoietic Stem Cell Transplantation; Malignant Hematological Diseases
Keywords: Umbilical Cord Blood Transplantation; Conditioning regimen
MeSH Terms: interventions — Cord Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 40 patients with malignant hematological diseases who underwent UCBT (Experimental)
  Interventions: Procedure: Umbilical Cord Blood Transplantation

INTERVENTIONS:
Procedure: Umbilical Cord Blood Transplantation — Compared with peripheral blood stem cell transplantation (PBST), UCBT has a higher transplantation rate, as cord blood stem cells are more primitive. Since the first successful umbilical cord blood transplantation (UCBT) in a child with severe Fanconi anemia reported by Gluckman et al. in France in 1988, cord blood has been widely used as a graft source of hematopoietic stem cells for the treatment of hematological diseases. The first sibling UCBT for leukemia was performed successfully by Professor Yongping Song in China, who played a pioneering role in the development of UCBT for leukemia in China. On the basis of previous research, the TFBC regimen (TBI/Flu/Bu/Cy) combined with UCBT is safe and feasible for the treatment of patients with high-risk malignant hematological diseases, which has enormous potential to improve patient outcomes.
  Other Names: Total Body Irradiation/Fludarabine/Busulfan/Cyclophosphamide

SUMMARY:
High-risk malignant hematological diseases refer to malignant hematological diseases, mainly include various types of leukemia, lymphoma, and multiple myeloma, with very poor prognoses, very short survival, and unsatisfactory outcomes.

Chemotherapy, hypomethylating agents (HMA), radiotherapy, targeted therapy, immunotherapy, and hematopoietic stem cell transplantation (HSCT) are common treatments for high-risk malignant hematological diseases. Because of the multiple lines and long duration of exposure to chemotherapy drugs in patients with high-risk malignant hematological diseases, monotherapy is inefficient, and radiotherapy is used frequently as an adjunct treatment to HSCT. Conventional myeloablative conditioning regimens before HSCT are comprised of cyclophosphamide/total body irradiation (Cy/TBI) and busulfan/cyclophosphamide (Bu/Cy). The reduced-toxicity myeloablative conditioning regimen, FBC, is the combination of Bu, Cy, and fludarabine (Flu), which has a strong immunosuppressive effect to ensure the success of engraftment of donor cells. Compared to the conventional intensified chemotherapy regimens, HMA have certain advantages of efficacy and safety and are the first-line treatment options for patients with acute myeloid leukemia (AML). Although monotherapy improves survival rate, the response rate is low. What's more, it is difficult to achieve sustained remission and long-term benefits. The current research hotspots are HMA combined with chemotherapy, targeted drugs such as BCL-2 inhibitors, immunotherapy, and cell therapy. Targeted therapy and immunotherapy are effective, but show a high prevalence of relapse, heavy treatment burden, and the need for long-term maintenance.

HSCT is an important therapy for the treatment of high-risk malignant hematological diseases, which could eliminate tumor cells through high-dose radiotherapy or chemotherapy, destroy the immune system of patients to prepare the engraftment of donor cells, and promote the reconstitution of hematopoiesis and immune recovery. HSCT has developed rapidly since the 1950s and has been performed in more than one million patients worldwide. HSCT is often the only definitive treatment available for patients with certain specific congenital or acquired diseases and is used in the treatment of many high-risk malignant hematological diseases. However, due to the strict criteria for HSCT, many patients do not have a matched donor. Since the first successful UCBT in a child with severe Fanconi anemia reported by Gluckman et al. in France in 1988, cord blood has been widely used as a graft source of hematopoietic stem cells for the treatment of hematological diseases.

Cord blood is rich in hematopoietic stem cells, endothelial progenitor cells, mesenchymal stem cells, and other stem/progenitor cells, as well as natural killer cells, Treg cells, and other immune cells, which have strong self-renewal and proliferation ability and low immunogenicity. The hematologic growth factors produced by these cells could act on the formation of myeloid cells and granulocytes, which are beneficial to hematopoietic reconstruction and recovery. It contains a variety of cytokines such as thrombopoietin, erythropoietin, stem cell factor, and multi-class interleukins. Some cytokines such as stem cell factor, IL-6, and IL-11 are much higher in cord blood than in peripheral blood. The potential mechanism by which UCBT exerts its therapeutic effect in patients with hematological diseases is largely the result of the interaction of multiple growth factors and stem/progenitor cells with the organism.

Compared with peripheral blood stem cell transplantation (PBST), UCBT has a higher transplantation rate, as cord blood stem cells are more primitive and purer than bone marrow stem cells. UCBT could be performed with four or more matches, and have a relatively lower rejection rate, lower relapse rate of malignant hematological diseases, and lower cumulative incidence of chronic graft-versus-host disease (GVHD), which greatly improves patient survival. Prof. Sun Zimin's team at Anhui Provincial Hospital was the first to use UCBT for the treatment of patients with AML and found that the cumulative incidence of chronic GVHD and relapse rate were significantly reduced.

Based on the above, the TFBC regimen (TBI/Flu/Bu/Cy) combined with UCBT is safe and feasible for the treatment of patients with high-risk malignant hematological diseases, which has enormous potential to improve patient outcomes. Therefore, we designed this clinical study on the TFBC regimen combined with UCBT for the treatment of high-risk malignant hematological patients to observe the impact on the engraftment rate, relapse rate, the cumulative incidence of GVHD, and survival.

DETAILED DESCRIPTION:
High-risk malignant hematological diseases are commonly seen in patients with advanced age, complex karyotypes, genes related to poor prognosis, failure to achieve remission after remission-inducing chemotherapy, and relapsed or refractory diseases.

The first sibling UCBT for leukemia was performed successfully by Professor Yongping Song in China, who played a pioneering role in the development of UCBT for leukemia in China.

In a retrospective study done by Prof. Sun Zimin's team, the efficacy of intravenous Bu/Cy versus TBI/Cy was compared in 331 patients from 8 centers who underwent single-unit umbilical cord blood transplantation (UCBT). It was reported that the cumulative incidence of neutrophil engraftment was higher in the TBI/Cy group than in the Bu/Cy group (98.0% versus 91.6%, P < 0.001), but the time to neutrophil engraftment was shorter in the Bu/Cy group than in the TBI/Cy group (16 days versus 19 days, P < 0.001). There was no significant difference in the non-relapse mortality, relapse rate, or survival rate between the two groups. What's more, the GVHD-free and relapse-free survival rate of patients was significantly increased, greatly improving patient survival. UCBT has also been widely used in other malignant hematological diseases such as acute lymphoblastic leukemia (ALL), lymphoma, and multiple myeloma. In 2017, UCBT was performed for the treatment of an adult AML patient at the Central Hospital of Wuhan, and the patient was successfully discharged from hospital. In 2020, UCBT was performed for the treatment of a 14-year-old patient with myelodysplastic syndrome at the Tai'an Central Hospital, and the patient achieved a good recovery with very mild rejection after transplantation and was finally discharged safely. Since the first successful UCBT in the Seventh Hospital of Zhongshan University in April 2021, 10 cases have been successfully performed, including an obese patient weighing 85 kg, a patient with strong positive panel reactive antibodies (PRA), and a patient with AML who received a second transplant after the first PBST. The overall success rate was 100% and the longest disease-free survival was 2 years. No patients died due to transplant-related mortality (TRM), only 1 case of severe GVHD occurred, and none of them underwent relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Gender is not limited, patients between 14 to 70 years old (including critical value);
2. High-risk malignant hematological diseases (acute lymphoblastic leukemia, acute/chronic myeloid leukemia, multiple myeloma, etc.) diagnosed by bone marrow aspiration or biopsy according to the WHO diagnostic criteria;
3. The indexes of cardiac function, liver and kidney function were within the following limits:(1) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3× Upper limit of normal (ULN); (2)Total bilirubin ≤ 3×ULN; (3) Serum creatinine ≤ 2×ULN or creatinine clearance ≥ 40mL/min; (4) Left ventricular ejection fraction (LVEF) as measured by echocardiography or multi-gated acquisition (MUGA) scan is within the normal range (> 50%);
4. Umbilical cord blood with HLA match ≥ 4/6;
5. Expected survival ≥3 months;
6. Karnofsky (KPS) score ≥60%, Eastern Tumor Cooperative group (ECOG) status ≤ 2;
7. Patient fully understood the nature of the study, and voluntarily participates and signs informed consent.

Exclusion Criteria:

1. Patients had serious adverse reactions to investigational drugs such as allergies;
2. Patients with a history of immunodeficiency, or other acquired or congenital diseases, immunodeficiency diseases, and a history of organ transplantation;
3. Patients with hypertension, ventricular arrhythmia requiring clinical intervention, acute coronary syndrome, congestive heart failure, stroke, or other grade III or higher cardiovascular events within 6 months;
4. Two or more surgeries were performed within 4 weeks prior to enrollment;
5. Patients with active viral infections, including HIV, HBV, HCV, TP;
6. Pregnant or lactating patients;
7. The patient is currently participating in another clinical studies;
8. Patients deemed unsuitable for inclusion by other investigators.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
The cumulative incidence of neutrophil engraftment and platelet engraftment | on day 28±7 following UCBT
  Neutrophil and platelet engraftment is defined as the first occurrence of 3 consecutive days with an absolute neutrophil count of at least 0.5×109/L and a platelet count of over 20×109/L for 7 consecutive days without transfusion support.
The time to reconstitution of hematopoiesis | on day 28±7 following UCBT
  Recovery of hemopoietic function after treatment
The cumulative incidence of transplant-related mortality (TRM) | within 100 days following UCBT
  Transplant-related mortality was defined as mortality due to any cause other than disease progression within 100 days of transplantation.

SECONDARY OUTCOMES:
The cumulative incidence and severity of pre-engraftment syndrome (PES) | on day 28±7 following UCBT
  Pre-engraftment syndrome (PES) is a condition occurring after umbilical cord blood transplantation (UCBT) characterized by fever and erythematous skin rash prior to neutrophil engraftment.
The cumulative incidence and grade of graft-versus-host disease (GVHD) | within 1 year following UCBT
  Graft-versus-host disease (GvHD) is a medical complication following the receipt of transplanted tissue from a genetically different person.
The cumulative incidence of relapse | within 1 year following UCBT
  We defined relapse as any clinical evidence of progression or recurrence of original diseases.
Overall survival rate | within 1 year following UCBT
  We estimated OS from the time of transplant until the date of death of any cause or last follow-up for patients still alive.
The cumulative incidence of adverse event | within 1 year following UCBT
  Following extraction of the tumor, a blood vessel burst causing increased blood loss during the procedure, an adverse event the surgeon did not expect.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow university, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Hu D, Yuan S, Zhong J, Liu Z, Wang Y, Liu L, Li J, Wen F, Liu J, Zhang J. Cellular senescence and hematological malignancies: From pathogenesis to therapeutics. Pharmacol Ther. 2021 Jul;223:107817. doi: 10.1016/j.pharmthera.2021.107817. Epub 2021 Feb 12. PMID 33587950
- [Background] Hellmich C, Moore JA, Bowles KM, Rushworth SA. Bone Marrow Senescence and the Microenvironment of Hematological Malignancies. Front Oncol. 2020 Feb 25;10:230. doi: 10.3389/fonc.2020.00230. eCollection 2020. PMID 32161723
- [Background] Auberger P, Tamburini-Bonnefoy J, Puissant A. Drug Resistance in Hematological Malignancies. Int J Mol Sci. 2020 Aug 24;21(17):6091. doi: 10.3390/ijms21176091. PMID 32847013
- [Background] Rambaldi A, Grassi A, Masciulli A, Boschini C, Mico MC, Busca A, Bruno B, Cavattoni I, Santarone S, Raimondi R, Montanari M, Milone G, Chiusolo P, Pastore D, Guidi S, Patriarca F, Risitano AM, Saporiti G, Pini M, Terruzzi E, Arcese W, Marotta G, Carella AM, Nagler A, Russo D, Corradini P, Alessandrino EP, Torelli GF, Scime R, Mordini N, Oldani E, Marfisi RM, Bacigalupo A, Bosi A. Busulfan plus cyclophosphamide versus busulfan plus fludarabine as a preparative regimen for allogeneic haemopoietic stem-cell transplantation in patients with acute myeloid leukaemia: an open-label, multicentre, randomised, phase 3 trial. Lancet Oncol. 2015 Nov;16(15):1525-1536. doi: 10.1016/S1470-2045(15)00200-4. Epub 2015 Sep 28. PMID 26429297
- [Background] Garcia-Manero G, Griffiths EA, Steensma DP, Roboz GJ, Wells R, McCloskey J, Odenike O, DeZern AE, Yee K, Busque L, O'Connell C, Michaelis LC, Brandwein J, Kantarjian H, Oganesian A, Azab M, Savona MR. Oral cedazuridine/decitabine for MDS and CMML: a phase 2 pharmacokinetic/pharmacodynamic randomized crossover study. Blood. 2020 Aug 6;136(6):674-683. doi: 10.1182/blood.2019004143. PMID 32285126
- [Background] Hu D, Gao YH, Yao XS, Gao H. Recent advances in dissecting the demethylation reactions in natural product biosynthesis. Curr Opin Chem Biol. 2020 Dec;59:47-53. doi: 10.1016/j.cbpa.2020.04.014. Epub 2020 May 24. PMID 32460136
- [Background] Aldea M, Andre F, Marabelle A, Dogan S, Barlesi F, Soria JC. Overcoming Resistance to Tumor-Targeted and Immune-Targeted Therapies. Cancer Discov. 2021 Apr;11(4):874-899. doi: 10.1158/2159-8290.CD-20-1638. PMID 33811122
- [Background] O'Donnell JS, Teng MWL, Smyth MJ. Cancer immunoediting and resistance to T cell-based immunotherapy. Nat Rev Clin Oncol. 2019 Mar;16(3):151-167. doi: 10.1038/s41571-018-0142-8. PMID 30523282
- [Background] Saad A, de Lima M, Anand S, Bhatt VR, Bookout R, Chen G, Couriel D, Di Stasi A, El-Jawahri A, Giralt S, Gutman J, Ho V, Horwitz M, Hsu J, Juckett M, Kharfan-Dabaja MA, Loren A, Meade J, Mielcarek M, Moreira J, Nakamura R, Nieto Y, Roddy J, Satyanarayana G, Schroeder M, Tan CR, Tzachanis D, Burn J, Pluchino L. Hematopoietic Cell Transplantation, Version 2.2020, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2020 May 1;18(5):599-634. doi: 10.6004/jnccn.2020.0021. PMID 32519831
- [Background] Yang G, Wang X, Huang S, Huang R, Wei J, Wang X, Zhang X. Generalist in allogeneic hematopoietic stem cell transplantation for MDS or AML: Epigenetic therapy. Front Immunol. 2022 Oct 4;13:1034438. doi: 10.3389/fimmu.2022.1034438. eCollection 2022. PMID 36268012
- [Background] Gluckman E, Broxmeyer HA, Auerbach AD, Friedman HS, Douglas GW, Devergie A, Esperou H, Thierry D, Socie G, Lehn P, et al. Hematopoietic reconstitution in a patient with Fanconi's anemia by means of umbilical-cord blood from an HLA-identical sibling. N Engl J Med. 1989 Oct 26;321(17):1174-8. doi: 10.1056/NEJM198910263211707. No abstract available. PMID 2571931
- [Background] Ehrhart J, Sanberg PR, Garbuzova-Davis S. Plasma derived from human umbilical cord blood: Potential cell-additive or cell-substitute therapeutic for neurodegenerative diseases. J Cell Mol Med. 2018 Dec;22(12):6157-6166. doi: 10.1111/jcmm.13898. Epub 2018 Oct 18. PMID 30334335
- [Background] Sun HP, Zhang X, Chen XH, Zhang C, Gao L, Feng YM, Peng XG, Gao L. Human umbilical cord blood-derived stromal cells are superior to human umbilical cord blood-derived mesenchymal stem cells in inducing myeloid lineage differentiation in vitro. Stem Cells Dev. 2012 Jun 10;21(9):1429-40. doi: 10.1089/scd.2011.0348. Epub 2011 Dec 5. PMID 22023173
- [Background] Sanchez-Petitto G, Rezvani K, Daher M, Rafei H, Kebriaei P, Shpall EJ, Olson A. Umbilical Cord Blood Transplantation: Connecting Its Origin to Its Future. Stem Cells Transl Med. 2023 Mar 3;12(2):55-71. doi: 10.1093/stcltm/szac086. PMID 36779789
- [Background] Zheng CC, Zhu XY, Tang BL, Zhang XH, Zhang L, Geng LQ, Liu HL, Sun ZM. Clinical separation of cGvHD and GvL and better GvHD-free/relapse-free survival (GRFS) after unrelated cord blood transplantation for AML. Bone Marrow Transplant. 2017 Jan;52(1):88-94. doi: 10.1038/bmt.2016.182. Epub 2016 Jul 4. PMID 27376453